CLINICAL TRIAL: NCT04234945
Title: Effect of Prophylactic Antibiotics for Hysterosalpingography on Post Procedure Morbidity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ahmadu Bello University Teaching Hospital (Other)
Responsible Party: Principal Investigator, Anisah Yahya, Dr, Ahmadu Bello University Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ABUTH Zaria
Record Dates: First submitted 2020-01-16; First posted 2020-01-21 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Infertility, Female; Pelvic Inflammatory Disease
MeSH Terms: conditions — Infertility, Female; Pelvic Inflammatory Disease | interventions — Doxycycline

STUDY DESIGN:
Intervention Model Description: Group A will be the study group and will be given oral Doxycycline capsule 100mg bd for 3/7. She will be instructed to commence the medication on day 7 of her next menstrual cycle and hysterosalpingogram will be done within the proliferative phase (Day 10) of the same menstrual cycle after cessation of bleeding.
  Group B will be the study group and will be given oral Multivitamin capsule i bd for 3/7. She will be instructed to commence the medication on day 7 of her next menstrual cycle and hysterosalpingogram will be done within the proliferative phase (Day 10) of the same menstrual cycle after cessation of bleeding
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The drugs given to participants in Groups A and B are in capsules and have thesame size and packaging but different colors. They will be put in a brown envelop to cover the color. The brown envelops will then be labelled with study number based in the numbers generated by the Random number table (WINPEPI) by a research assistant to ensure the principal investigators do not know the drug inside the brown envelopes. The participants will take the drugs at home. This ensures that the care provider, investigators and outcomes assessors do not know the drug the patient takes. However the patient will know the drug she takes since the drug is labelled.
  The
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study (Experimental): Group A will be the study group and will be given oral Doxycycline capsule 100mg bd for 3/7.
  Interventions: Drug: Doxycycline Capsule
- control (Placebo Comparator): Group B will be the study group and will be given oral Multivitamin capsule i bd for 3/7
  Interventions: Drug: Multivitamins W/Iron Tab

INTERVENTIONS:
Drug: Doxycycline Capsule — Group A will be the study group and will be given oral Doxycycline capsule 100mg bd for 3/7. She will be instructed to commence the medication on day 7 of her next menstrual cycle and hysterosalpingogram will be done within the proliferative phase (Day 10) of the same menstrual cycle after cessation of bleeding.
  Other Names: Doxycap. Registration No: MAL 19921000A
  Arms: study
Drug: Multivitamins W/Iron Tab — Group B will be the study group and will be given oral Multivitamin capsule i bd for 3/7. She will be instructed to commence the medication on day 7 of her next menstrual cycle and hysterosalpingogram will be done within the proliferative phase (Day 10) of the same menstrual cycle after cessation of bleeding
  Other Names: Haemaron
  Arms: control

SUMMARY:
The study will be a parallel randomised trial. There are two groups. The first group will be given prophylactic antibiotics before a procedure (hysterosalpingography) and the second group will be given a placebo(multivitamin). Outcomes will then be assessed.

DETAILED DESCRIPTION:
Hysterosalpingography is a radiological procedure that outlines the female genital tract1. It is routinely done as part of work up for female infertility with the aim of identifying lesions that may cause female factor infertility1. It is considered as a minor gynaecological procedure2.

The procedure involves exposing the cervix with a bivalve speculum and injecting a contrast medium through a cannula that is applied to the cervix. Images of the genital tract are then obtained by fluoroscopy.

The lower genital tract is rich in micro flora. The natural milieu of the lower genital tract prevents infection. However, the upper genital tract is sterile. Microorganisms can ascend from the lower genital tract to the upper genital tract through the cervix and lead to infections. Infections of the upper genital tract can result in acute or chronic pelvic infection with subsequent chronic abdominal pain, ectopic pregnancy, menstrual irregularities and infertility as a result of inflammation and scarring of the fallopian tubes.

Hysterosalpingography can lead to transcervical transmission of microorganisms from the lower genital tract to the upper genital tract. Cervical trauma during the procedure can facilitate ascending infection. Also, direct transcervical transfer of microorganisms from the lower genital tract to the upper genital tract can occur.

Different approaches of preventing iatrogenic upper genital tract infection following hysterosalpingography exist. Prophylactic antibiotics can be given to all clients undergoing the procedure. On the other hand, prophylactic antibiotics may be limited to only those that have symptoms suggestive of genital tract infection based on their history. However, this may not suffice because some genital tract infections are mainly asymptomatic. Another approach is to screen all clients undergoing hysterosalpingography for genital tract infection and treat as necessary. Screening may also be limited to those with history suggestive of genital tract infection. This approach may also miss the clients with asymptomatic infections.

Despite the possibility of iatrogenic upper genital tract infection following hysterosalpingography and availability of possible approaches in preventing such infection, there is no standard recommendation for the use of prophylactic antibiotics for hysterosalpingography2,3.

Thinkhamrop et al conducted a review on prophylactic antibiotic for transcervical intrauterine procedures2. The procedures included the collection of endometrial tissue to assess the cause of abnormal uterine bleeding, hysterosalpingography for infertility evaluation, hysteroscopy for intrauterine cavity diagnosis and treatment, and the evacuation of conceptive products. They reported that there were no available randomized controlled trials on the subject matter to enable recommendations for the use of antibiotics for such procedures.

This study aims at determining the effect of prophylactic antibiotic for Hysterosalpingography on post procedure morbidity. Specific objectives include determining the effect of prophylactic antibiotic for hysterosalpingography on post procedure febrile morbidity, infectious morbidity and need for antibiotic therapy. Effect on adverse effect of the antibiotics will also be reported.

METHODOLOGY STUDY DESIGN The study will be a randomized controlled trial. STUDY AREA The study will be conducted at the departments of Obstetrics and Gynaecology and radiology Ahmadu Bello University Teaching Hospital, Zaria.

The participants will be recruited from the departments of Obstetrics and Gynaecology and radiology, Ahmadu Bello University Teaching Hospital, Zaria, as they present for review and work up for infertility.

Patients will be followed up for the outcome via mobile calls and outpatient gynaecology clinic attendance.

STUDY POPULATION The study will comprise of women who present to the department of radiology Ahmadu Bello University Teaching Hospital, Zaria for hysterosalpingography as part of routine work up for infertility.

SAMPLING APPROACH/RANDOMISATION A probability sampling method will be used. Simple random sampling using a computer generated table of random numbers will be used. The WINPEPI version 11.65 software was used to generate the table of random numbers. The numbers 001-156 will be randomly allocated to two groups A and B. Group A will be the study group and group B will be the control group (see appendix). Each number from the table of random numbers will be copied on separate paper and then sealed in a brown envelope. The envelopes will then be kept inside a box after shuffling.

Each patient will be allocated to the group that the number she picks corresponds to on the computer printout.

SAMPLE SIZE DETERMINATION:

The sample size for each group was determined by using the statistical formula for comparison of proportions. Each group will be rounded up to 78.

SAMPLING RECRUITEMENT:

Women that fulfil the inclusion criteria will be counselled about the study in the departments of Obstetrics and Gynaecology.

After obtaining a written consent, the consent form will be attached to the radiology request form for hysterosalpingography and they will be referred to the radiology departments.

At the radiology departments, participants will be requested to pick one of the brown envelopes which will contain the randomization group.

Group A will be the study group and will be given oral Doxycycline capsule 100mg bd for 5/7. She will be instructed to commence the medication on day 1 of her next menstrual cycle and hysterosalpingogram will be done within the proliferative phase of the same menstrual cycle after cessation of bleeding.

Group B will be given oral multivitamin capsule i bd for 5/7. She will be instructed to commence the medication on day 1 of her next menstrual cycle and hysterosalpingogram will be done within the proliferative phase of the same menstrual cycle after cessation of bleeding.

The clients will be contacted over the phone for follow up 24 hours after the procedure. They will also be requested to present to the emergency gynaecology unit in case they develop any symptom. All clients will be booked for routine follow up appointment in the gynaecology clinic two weeks after the procedure. The clients will also be given digital thermometers and taught how to use them in case they develop fever before they present to the emergency unit.

DATA COLLECTION METHOD:

A proforma will be filled for the participants. This will include Biodata, contact, details of their Sociodemographic and reproductive profiles. History of previous minor gynaecological procedures will also be obtained.

ANALYTICAL APPROACH Data will be analysed using the statistical package for social sciences (SPSS) version 20.0. Chi-square test will be used to analyse categorical data and student t-test will be used to analyze continuous data. Logistic regression will be used to examine the influence of compounders. A p- value of less than 0.05 will be considered as significant.

The primary and secondary outcomes will be analysed to determine any significant statistical differences. A p-value of less than 0.05 will be considered as significant. Relative risk (95% confidence level) will also be determined for every outcome.

The socio-demographic characteristics, reproductive profile and history of previous minor gynaecological procedure will be analysed to determine whether there are any significant differences within the two groups which may affect the outcome of the study. Chi-square test will be used for categorical data and student t-test will be used for continuous data.

If there is statistically significant difference in the characteristics of the participants, logistic regression will be used to eliminate the effect of these differences on the outcome of the study.

ELIGIBILITY:
Inclusion Criteria:

* Women who present for hysterosalpingography as routine work up for infertility.

Exclusion Criteria:

* Women who present for hysterosalpingography for other indications apart from infertility.
* Women with history of use of antibiotics within two weeks of the procedure.
* Women with symptoms of acute pelvic infection

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — self representation
Enrollment: 78 (Estimated)
Dates: Start 2020-01-13 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
No of participants in each arm that develop Fever | 24 hours to 10 days after the procedure
  Axillary temperature of ≥38.0oC
No of participants in each arm that develop Clinical features of pelvic infection | within 2 weeks of the procedure
  Lower abdominal pain, abnormal vaginal discharge, radiological/laboratory evidence of pelvic infection ( Significant fluid collection in the pouch of Douglas)
No of participants in each arm that develop the Need for antibiotics treatment. | within 2 weeks of procedure
  Requirement for antibiotic therapy for pelvic infection

SECONDARY OUTCOMES:
No of participants in each arm that develop Side effects to the antibiotics | within 24 hours after the procedure.
  Nausea, vomiting, Diarrhea, skin reaction

CONTACTS AND LOCATIONS:
Overall Officials: Anisah Yahya, MBBS, Principal Investigator — Ahmadu Bello University
Locations (1):
- Ahmadu Bello University Teaching Hospital Shika-Zaria, Zaria, Kaduna State, Nigeria

IPD SHARING:
Plan to Share IPD: No